CLINICAL TRIAL: NCT03181711
Title: A Comparison Between DIAGNOcam and Bitewing Radiographs as Diagnostic Methods for Approximal Caries in Primary Teeth.
Brief Title: Is DIAGNOcam Comparable to Bitewing Radiographs as a Diagnostic Method for Approximal Caries in Primary Teeth?
Acronym: Diagncamera
Status: Completed | Type: Observational
Sponsor: Malmö University (Other)
Responsible Party: Principal Investigator, Susanne Brogårdh-Roth, Principle Investigator, Malmö University
Other Study IDs: DIAGNOcam Malmo U
Record Dates: First submitted 2017-06-04; First posted 2017-06-09 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Caries
Keywords: Dental caries; Tooth, deciduous; Children; Radiography/bitewing; diagnostic imaging
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
BACKGROUND: To diagnose caries in clinical practice today, a combination of clinical examination with mirror and probe, and in sometimes x-ray images are used. For surfaces in contact with other teeth X-rays (preferably bitewing) are often required. Even though the radiation doses in bitewings are small, it is important to weigh risks against the benefit to avoid unnecessary radiation.

There are other methods for diagnosing caries based on different forms of laser light. One such technique is based on the translucency of the teeth. The light is within the near infrared light (NIR) area. A product named DAIGNOcam (diagnostic camera) is using this technology. The light is led in a hand piece held against the tooth. The tooth is illuminated and the caries lesions can be seen like dark spots on a computer monitor screen. The technique is mainly used in adult patients and permanent teeth. However, there is no complete evaluation of how well the technology diagnoses caries in milk teeth. From a radiation hygiene point of view, it is particularly important to reduce the amount of X-rays to young individuals. X-rays are often experienced as difficult by younger children, which leads to poorer diagnostics. It is important to identify early caries in milk teeth as these teeth have thinner enamel and a more "porous" dentin. This may lead to that caries progress much faster thus more difficult to fix. This in turn leads to a risk of toothache and that the damage becomes so extensive that the tooth must be removed.

OBJECTIVE: To investigate diagnostic accuracy / precision in caries diagnosis between teeth using DIAGNOcam in milk teeth comparable to caries diagnostics using bitewing x-rays.

RESEARCH QUESTIONS:

* Is DIAGNOcam a reliable diagnostic method for diagnosing caries in between teeth (approximal caries) in milk teeth?
* How does child experience caries diagnosing performed with DIAGNOcam compared to X-rays? INVESTIGATION VARIABLES: Caries data are recorded according to the accepted diagnostic method at the surface level. Each examined tooth surface is assessed as either 1) intact; 2) caries only in enamel; 3) caries i dentin; or 4) the surface can not be judged. The same classification is used for X-rays and DIAGNOcam.

The children will also be able to rate their experience of the X-ray examination and the DIAGNOcam survey using a Faces pain scale to see if there is any difference in experience between the different methods of investigation.

DETAILED DESCRIPTION:
BACKGROUND: Caries is a multifactorial and infectious disease. To diagnose caries in clinical practice, a combination of clinical examination with mirror and probe (visual-tactile examination) is used today, as well as in some cases standardized x-rays called bitewing x-ray (bw). Visual-tactile examination is enough to diagnose caries on buccal and lingual/palate surfaces. However, for approximal surfaces, X-rays are often required to ensure diagnosis and to assess the spread of a caries lesion in the tooth. Bitewing X-rays are the single best diagnostic tools for diagnosing caries in approximal surfaces. An X-ray examination should always be performed on individual indications. At bw the radiation doses are small. Nevertheless, it is important to weigh risks against the benefit to avoid unnecessary radiation. Reducing the number of dental radiographs is also important from the perspective of safe dental care where one strives to make use of and not harm.

There are other methods for diagnosing caries based on different forms of laser light that can detect caries. Previously, these techniques have only been used for occlusal surfaces and buccal/lingual/palate tooth surfaces, not for diagnostics between teeth. For some time now, the translucency of the teeth is used in a technique. The light is within the so-called NIR area - near infrared light (non-wavelength wavelength). On the market, a product (DAIGNOcam) uses this technology. The light is led in a hand piece (like a little bigger pen) held against the tooth, one tooth at a time. The tooth is illuminated and a digital video camera on the hand piece projects a computer monitor image. In the picture, the caries lesions are seen like dark spots. These correspond to a qualitative defect in the enamel or dentin, i.e. an area where various minerals were lost / dissolved due to caries (demineralized area). The image can be saved in the patient's dental record in the same way as regular photos or X-rays. DIAGNOcam provides a qualitative response - one looks primarily if it is caries or not. It will then be a supplement to the usual survey with mirror and probe. The technique is mainly used in adult patients and permanent teeth. DIAGNOcam is currently available in clinical practice since a number of years. However, there is no complete evaluation of how well the technology diagnoses caries in primary teeth. This is unfortunate for mainly two reasons: from a radiation hygiene point of view, it is especially important to reduce the amount of X-rays to young individuals; Intra-oral X-rays are often experienced as difficult to manage by younger children, which leads to poorer diagnostics. It is important to identify early caries lesions in primary teeth as these teeth have a thinner enamel and a less mineralized dentin, which causes a caries lesion to progress much faster. This may lead to difficulties in restoring the teeth as well as pain from pulpal involvement. If the carious lesion is extensive, this may lead to tooth extraction.

OBJECTIVE: To investigate diagnostic accuracy / precision in caries diagnostics using DIAGNOcam in primary teeth comparable to caries diagnostics using bitewing x-rays.

PRIMARY RESEARCH QUESTION:

• Is DIAGNOcam a reliable diagnostic method for diagnosing approximal caries in primary teeth?

SECONDARY RESEARCH QUESTION:

• How does children experience caries diagnosing performed with DIAGNOcam compared to X-rays? INVESTIGATION VARIABLES: Caries data are recorded according to the standardized diagnostic method at surface level (dental sites with approximal contacts). Each examined tooth surface is assessed as either 1) intact; 2) caries only in enamel; 3) caries i dentin; or 4) the surface cannot be judged. The same classification is used for X-rays and DIAGNOcam.

The children will also be able to rate their experience of the X-ray examination and the DIAGNOcam survey using a Faces pain scale to see if there is any difference in experience between the different methods of investigation.

KNOWLEDGE GAINS: New methods should always be evaluated before implementation to ensure good care. There are no evaluated diagnostic methods that do not use ionised radiation (X-ray) for caries diagnosing of approximal surfaces in contact with another tooth. If DIAGNOcam in evaluation shows the same diagnostic accuracy as X-ray, this may reduce the use of dental x-ray for children. If DIAGNOcam is found to have poorer diagnostic accuracy, the method should be avoided as a caries diagnostic method in primary teeth. The latter is based on the fact that children should not be exposed to unnecessary examinations or interventions that do not result in health benefits.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 4-8
* Radiograph bitewings not older than 3 months
* First and second primary mandibular or maxillary molars present
* Parental consent

Exclusion Criteria:

* Children not in need of bitewing radiographs
* Children with mineralization disturbances, chronic diseases, functional or psychological disabilities that influence the possibility to participate
* Children who of other reasons have difficulties to participate

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 50 patients who meet the inclusion criteria are recruited consecutively at the dep of pediatric dentistry, Faculty of Odontology in Malmö. In order to obtain a spread in caries, there are no restraints regarding dental health in the children. It is important to include both children with a lot of caries and children with little or even no caries.
  No power calculation can be performed as there is no basis for obtaining the size of the study population. However, there are similar studies on other diagnostic methods in which diagnostic reliability was investigated with a study material of 50 patients. Therefore, the study intends to include 50 patients resulting in at least 400 surfaces.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
number of surfaces with manifest approximal caries lesions | measured at the dental examination
  approximal caries in primary molars registered in radiographs (bitewings) or with DIAGNOcam. Caries lesions clearly visible in dentin.

SECONDARY OUTCOMES:
Children´s perception of pain during examination with radiographs (bitewings) and DIAGNOcam. | measured at the dental examination
  Child assessment of pain using Facial Pain Scale

CONTACTS AND LOCATIONS:
Overall Officials: Susanne I Brogårdh-Roth, Doctor, Principal Investigator — Malmö University
Locations (1):
- Malmö University, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- Available data/document: Study Protocol — http://mah.se — can be requested by mail Karin.Ridell@mah.se